CLINICAL TRIAL: NCT04451811
Title: A Pharmacokinetic Dose Proportionality Study of OPL-002 in Healthy Volunteers
Brief Title: A PK Dose Proportionality Study of OPL-002 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oppilan Pharma Ltd (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OPL-002-102
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OPL-002 SDD 20 mg (Experimental): 20 mg SDD formulation of OPL-002
  Interventions: Drug: OPL-002
- OPL-002 5 mg Tablet (Experimental): 5 mg tablet formulation of OPL-002
  Interventions: Drug: OPL-002
- OPL-002 20 mg Tablet (Experimental): 20 mg tablet formulation of OPL-002
  Interventions: Drug: OPL-002

INTERVENTIONS:
Drug: OPL-002 — Spray dried dispersion and tablet formulation

SUMMARY:
This is a single center, randomized, open-label, three-way crossover, single dose, pharmacokinetic dose proportionality study of oral OPL-002 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (of non-childbearing potential only) between 18 and 55 years of age.
* Females must be of non-childbearing potential and must have undergone one of the following sterilization procedures, and have official documentation, at least 6 months prior to the first dose:

  1. hysteroscopic sterilization;
  2. bilateral tubal ligation or bilateral salpingectomy;
  3. hysterectomy;
  4. bilateral oophorectomy, or;
  5. be postmenopausal with amenorrhea for at least 1 year prior to the first dose and have FSH serum levels consistent with postmenopausal status as per investigator judgment.
* Male subjects must use reliable forms of contraception from screening to 30 days after the end of dosing.
* Good general health as determined by medical history, and by results of physical examination, vital signs, ECG, and clinical laboratory tests obtained within 28 days (4 weeks) prior to study drug administration.

Exclusion Criteria:

* History or presence of any clinically significant organ system disease that could interfere with the objectives of the study or the safety of the subjects.
* pressure and heart rate are outside the ranges 90-140 mmHg systolic, 40-90 mmHg diastolic, heart rate 60-100 beats/min.
* 12-lead ECG with any abnormality judged by the Investigator to be clinically significant, QRS >= 110 milliseconds (msec), QT/QTcF interval of > 450 msec for men or >470 msec for women, or PR > 200 msec.
* Presence or history of any abnormality or illness, which in the opinion of the Investigator may affect absorption, distribution, metabolism or elimination of the study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
AUC of OPL-002 | 0 to 48 hours

SECONDARY OUTCOMES:
Dose proportionality of 5 and 20 mg | 0 to 48 hours
Absolute lymphocyte count | 0 to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gregg, MD, Study Director — Oppilan Pharma Ltd
Locations (1):
- Celerion, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No